CLINICAL TRIAL: NCT03636308
Title: Phase II Trial Comparing Nab-paclitaxel Plus S-1 Versus Nab-paclitaxel Plus Gemcitabine in First-line Treatment of Patients With Advanced Pancreatic Cancer
Brief Title: Nab-paclitaxel Plus S-1(AS) Versus Nab-paclitaxel Plus Gemcitabine(AG) in Patients With Advanced Pancreatic Cancer
Acronym: ASAGPAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASAG01
Record Dates: First submitted 2018-08-01; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Pancreatic Cancer
Keywords: advanced pancreatic cancer; nanoparticle albumin-bound paclitaxel; S-1; gemcitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Taxes; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; S 1 (combination); Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AS：Nanoparticle albumin-bound paclitaxel，S-1 (Experimental): Nanoparticle albumin-bound paclitaxel is given at 125 mg/m2 intravenously on day 1 of each 14 day cycle.
  S-1 is orally administered (BSA<1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2, 50mg bid, BSA>1.5m2, 60mg bid) on day 1-7 of each 14 day cycle.
  Interventions: Drug: nanoparticle albumin-bound paclitaxel; Drug: S1
- AG：Nanoparticle albumin-bound paclitaxel，Gemcitabine (Active Comparator): Nanoparticle albumin-bound paclitaxel is given at 125 mg/m2 intravenously on day 1 and 8 of each 21 day cycle.
  Gemcitabine is given at 1000mg/m2 intravenously on day 1 and 8 of each 21 day cycle.
  Interventions: Drug: nanoparticle albumin-bound paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: nanoparticle albumin-bound paclitaxel — Nanoparticle albumin-bound paclitaxel is given at 125 mg/m2 intravenously on day 1 of each 14 day cycle or day 1 and 8 of 21 day cycle.
  Other Names: nab-paclitaxel; Abraxane; ABI-007
Drug: S1 — S-1 is orally administered (BSA<1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2, 50mg bid, BSA>1.5m2, 60mg bid) on day 1-7 of each 14 day cycle.
  Arms: AS：Nanoparticle albumin-bound paclitaxel，S-1
Drug: Gemcitabine — Gemcitabine is given at 1000mg/m2 intravenously on d1 and 8 of each 21 day cycle.
  Arms: AG：Nanoparticle albumin-bound paclitaxel，Gemcitabine

SUMMARY:
This is a randomized phase II trial comparing the first-line treatment with nab-paclitaxel plus S-1(AS) and nab-paclitaxel plus gemcitabine(AG) in advanced pancreatic ductal adenocarcinoma (PDA) with primary tumor nonexcision in Chinese patients.

DETAILED DESCRIPTION:
Advanced pancreatic ductal adenocarcinoma (PDAC) is an aggressive and chemo-resistant disease with extremely low 5-year survival rate. Gemcitabine has been the cornerstone of metastatic PDAC treatment for more than a decade , although survival benefit was very poor. Nab-paclitaxel added to gemcitabine has showed improving survival and overall response rate vs gemcitabine alone in metastatic PDAC first-line treatment in the MPACT phaseIII study, which represents one of the standards of care in advanced PDAC therapy. S-1 is an oral 5-fluorouracil (5-FU) prodrug, and shown to be non-inferior to gemcitabine on OS for unresectable pancreatic cancer. Meanwhile, adjuvant chemotherapy with S-1 monotherapy was found to significant prolong survival of pancreatic cancer patients when compared with gemcitabine. This study is to explore the efficacy and safety of nab-paclitaxel plus S-1(AS) and nab-paclitaxel plus gemcitabine(AG) as first-line treatment in advanced pancreatic ductal adenocarcinoma (PDA) with primary tumor nonexcision in Chinese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed-consent form.
2. Age no less than 18 years.
3. Histologically confirmed locally advanced or metastatic pancreatic ductal adenocarcinoma, with RECIST measurable lesions.
4. Eastern Cooperative Oncology Group (ECOG) 0-1 with life expectation of no less than 12 weeks.
5. Patients must have received no previous chemotherapy or investigational therapy for the treatment of locally advanced or metastatic disease.
6. At least 4 weeks since completion of the last operation except for diagnostic biopsy.
7. At least 4 weeks since completion of radiotherapy to lesions.
8. Not suitable for local treatment.
9. Adequate liver/bone marrow function.
10. Human Chorionic Gonadotropin (HCG) test negative for female with contraception measure until 3 months after study end.
11. Compliant, and can be followed up regularly.

Exclusion Criteria:

1. Received chemotherapy or investigational therapy for the treatment of locally advanced or metastatic disease.
2. Pregnant or breast-feeding female, or not willing to take contraception measures during study.
3. Serious infection requiring antibiotics intervention during recruitment.
4. Allergic to study drug.
5. More than grade 1 neuropathy.
6. Uncontrolled brain metastasis or mental illness.
7. Congestive heart failure, uncontrolled cardiac arrhythmia, etc.
8. Other malignancy within 5 years.
9. Can't be followed up or obey protocol.
10. Ineligible by the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST)(every 3 cycles in AS or every 2 cycles in AG).

SECONDARY OUTCOMES:
Objective response rate of primary tumor | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST)(every 3 cycles in AS or every 2 cycles in AG).
Progression-free survival | up to 15 months
  Measure of time from study treatment to disease progression or death.
Overall survival | up to 2 years
  Measure of time from study treatment to patient's death or lost to follow-up.
Disease control rate | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The sum of rates of partial response, complete response and steady disease based on Response Evaluation Criteria In Solid Tumors (RECIST).
The incidence of treatment related emergent adverse events（Safety and Tolerance） | Until 28 days after the deadline of enrollment
  Adverse reactions evaluation is based on the National Cancer Institute adverse event General terminology Standard [CTCAE] 4.0 version

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Professor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin M, Liu HL, Xue J, Ma H, Liu JL, Lin ZY, Wang J, Bao LQ, Luo ZG, Yu XJ, Li S, Hu JL, Zhang T. Nab-paclitaxel plus S-1 versus nab-paclitaxel plus gemcitabine in patients with advanced pancreatic cancer: a multicenter, randomized, phase II study. Oncologist. 2024 Oct 3;29(10):e1406-e1418. doi: 10.1093/oncolo/oyae171. PMID 38990195
- [Derived] Zong Y, Yuan J, Peng Z, Lu M, Wang X, Shen L, Zhou J. Nab-paclitaxel plus S-1 versus nab-paclitaxel plus gemcitabine as first-line chemotherapy in patients with advanced pancreatic ductal adenocarcinoma: a randomized study. J Cancer Res Clin Oncol. 2021 May;147(5):1529-1536. doi: 10.1007/s00432-020-03442-0. Epub 2020 Nov 15. PMID 33191450